CLINICAL TRIAL: NCT01838369
Title: A Single-arm, Open-label, Phase 2 Clinical Trial Evaluating Disease Response Following Treatment With BI-505, a Human Anti-Intercellular Adhesion Molecule 1 Monoclonal Antibody, In Patients With Smoldering Multiple Myeloma
Brief Title: A Phase II Study of BI-505 in Smoldering Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-BI-505-02
Record Dates: First submitted 2013-03-26; First posted 2013-04-24 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2015-05

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BI-505 (Experimental)
  Interventions: Drug: BI-505

INTERVENTIONS:
Drug: BI-505

SUMMARY:
The purpose of this study is to investigate the effect of BI-505 on tumor burden in patients diagnosed with smoldering multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Smoldering multiple myeloma based on the International Myeloma Working Group criteria:

  * Serum M-protein greater than or equal to 3 g/dL and/or bone marrow plasma cells greater than or equal to 10 percent.
  * Absence of end-organ damage such as lytic bone lesions, anemia, hypercalcemia or renal failure that can be attributed to a plasma cell proliferative disorder.
* Male or female, 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1.

Exclusion Criteria:

* Patients with a diagnosis of symptomatic multiple myeloma or a clinical suspicion of an ongoing progression into symptomatic multiple myeloma.
* Prior or current treatment having a proven or potential impact on myeloma cell proliferation or survival (including conventional chemotherapies, biological therapies, immunomodulatory drugs, or proteasome inhibitors), as judged by the Investigator.
* Severe other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess the change in disease activity measured as M-protein levels in serum/urine following BI-505 treatment compared to base line according to the International Myeloma Working Group (IMWG) uniform response criteria | M-protein will be measured at screening, prior to each dose and at end of study visit, for up to 19 weeks.

SECONDARY OUTCOMES:
The clinical safety of BI-505 will be assessed by reporting the numbers of AEs, the severity and the relationship to IMP. | At each visit and up to 28 days after the last dose.
  Safety will be assessed by measuring the following clinical safety parameters; Adverse events, vital signs, clinical laboratory tests, ECG and immunogenicity.
The pharmacokinetic profile of BI-505 will be determined by calculating the following pharmacokinetic parameters: AUC, % AUCex, Cmax, Tmax, CL, Vss and T1/2. | Up to 28 days after the last dose.
The pharmacodynamics of BI-505 will be assessed by measuring soluble biomarkers and ICAM-1 saturation on bone marrow plasma cells. | Up to 28 days after the last dose.
The immunogenicity profile of BI-505 will be assessed by measuring antibodies towards BI-505. | Prior to first dose and at 28 days after the final dose.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hansson, MD, PhD, Principal Investigator — Department of Hematology,Skåne University Hospital
Locations (1):
- Department of Hemtaology, Skåne University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Wichert S, Juliusson G, Johansson A, Sonesson E, Teige I, Wickenberg AT, Frendeus B, Korsgren M, Hansson M. A single-arm, open-label, phase 2 clinical trial evaluating disease response following treatment with BI-505, a human anti-intercellular adhesion molecule-1 monoclonal antibody, in patients with smoldering multiple myeloma. PLoS One. 2017 Feb 3;12(2):e0171205. doi: 10.1371/journal.pone.0171205. eCollection 2017. PMID 28158311